CLINICAL TRIAL: NCT00792922
Title: Research to Programs for Trachoma Elimination: Antibiotic Trial
Brief Title: Partnership for Rapid Elimination of Trachoma
Acronym: PRET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00018439
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Trachoma
Keywords: Trachoma; Azithromycin; Mass treatment
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: The study was a factorial study model to begin with in all 3 countries (Niger,Tanzania and Gambia) but because we never stopped treatment in Tanzania and Niger site.Hence the study design was collapsed to a simple design in Tanzania and Niger.The study model was kept as a factorial design for the Gambia site.
  Protocol Enrollment refers to the number of communities, not the number of participants enrolled.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ≥90% coverage with azithromycin target (Active Comparator): Selected communities will receive mass treatment annually for three years.
  Interventions: Drug: Azithromycin
- 80%-89% coverage with azithromycin target (Active Comparator): Selected communities will receive mass treatment annually for three years.
  Interventions: Drug: Azithromycin
- ≥90% coverage with azithromycin , treatment based (Active Comparator): Treatment to be administered at baseline then continued yearly if trachoma prevalence is greater than 5%
  In Niger, treatment will be every 6-months for children ages twelve and under.
  Interventions: Drug: Azithromycin
- 80%-89% coverage with azithromycin : treatment based (Active Comparator): Treatment to be administered at baseline then continued yearly if trachoma prevalence is greater than 5%
  In Niger, treatment will be every 6-months for children ages twelve and under.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Comparison of community coverage rate
  Other Names: Zithromax
  Arms: 80%-89% coverage with azithromycin target; ≥90% coverage with azithromycin target
Drug: Azithromycin — Comparison of coverage levels at baseline treatment followed by annual treatment if prevalence of trachoma is >5%. In Niger, there will be a comparison of coverage levels in everyone versus in children ages twelve and under who are treated every 6-months.
  Other Names: Zithromax
  Arms: 80%-89% coverage with azithromycin : treatment based; ≥90% coverage with azithromycin , treatment based

SUMMARY:
Trachoma, an ocular infection caused by C. trachomatis, is the second leading infectious cause of blindness worldwide. Years of repeated infection with C. trachomatis cause the eyelid to scar and contract and ultimately to rotate inward such that the eyelashes rub against the eyeball and abrade the cornea (trichiasis). The World Health Organization (WHO) has endorsed a multi-faceted strategy to combat trachoma, which includes the use of antibiotic treatment to reduce the community pool of infection with C. trachomatis. The objective of this study is to conduct a randomized, community-based trial in three countries (Niger, Tanzania and The Gambia), representing different baseline endemicities, of alternative coverages and frequencies of administration of mass antibiotic treatment as well as to determine the cost-effectiveness of these different strategies from a program perspective.

DETAILED DESCRIPTION:
A randomized, 2x2 factorial designed trial will be implemented in each of the three countries. Communities will be randomized to two different coverage targets (80%-89% versus ≥90%) for three years of mass treatment.

In The Gambia and Tanzania, communities will be further randomized to yearly mass treatment versus mass treatment at baseline followed by yearly mass treatment only if trachoma prevalence in sentinel children is greater than 5%. The communities will continue to be followed and treatment will resume if trachoma prevalence is found to be 20% or greater at the 12 or 18 month surveys.

In Niger, communities will be randomized to the different coverage levels for annual mass azithromycin distribution and further randomized to biannual treatment at the two coverage targets for children ages twelve or younger.

Cross-sectional rates of trachoma and infection will be determined by examining sentinel children, age five years or younger, randomly selected from each community based on a community census. The census will be updated each year, and villages will be monitored at baseline, 6, 12, 18, 24, 30, and 36 months for infection and clinical disease.

The three-year study is in accord with the WHO guidelines which recommend three years of annual mass treatment followed by a re-survey to determine need for further treatment. The investigators will evaluate the efficacy of guiding further mass treatment according to a laboratory test for Chlamydia or WHO guidelines. Where investigators estimate communities have infection rates less than 5% in sentinel children, or trachomatous inflammation (TF) ( rates less than 5%, the community will be "graduated" from further mass treatment and followed for up to three years to look for evidence of re-emergent infection and disease. If rates of infection are found to be 20% or more return at the 12 or 18 month survey, mass treatment will be re-initiated.

ELIGIBILITY:
Inclusion criteria for communities:

* Communities are located in the target districts and accessible by vehicle
* The community leaders consent to have the community enrolled
* Rapid assessment and/or available data suggest trachoma rates are higher than 20% in the community.
* The community size is <5,000 persons or >250 persons.

If a community meets the inclusion criteria and community leaders consent to have the community enrolled, then sentinel children will be selected based on the following criteria:

* The child is age 5 years or younger
* The child must be a resident in an eligible, sample community (defined as either living in the community since birth, or moved in with parents or guardians).
* The child must not have an ocular condition that would preclude grading trachoma or taking an ocular specimen.
* The child must be willing to have a swab taken as part of being a sentinel child (this is critical for The Gambia and Tanzania, as each swab result counts towards meeting the stopping rule)
* The child must have an identifiable guardian capable of providing consent to participate.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2008-05; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila West, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (2):
  - UCSF Proctor Foundation, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
- London School of Hygiene and Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldenburg CE, Amza A, Cooley G, Kadri B, Nassirou B, Arnold BF, Rosenthal PJ, O'Brien KS, West SK, Bailey RL, Porco TC, Keenan JD, Lietman TM, Martin DL. Biannual versus annual mass azithromycin distribution and malaria seroepidemiology among preschool children in Niger: a sub-study of a cluster randomized trial. Malar J. 2019 Dec 3;18(1):389. doi: 10.1186/s12936-019-3033-2. PMID 31796025
- [Derived] Kim JS, Oldenburg CE, Cooley G, Amza A, Kadri B, Nassirou B, Cotter SY, Stoller NE, West SK, Bailey RL, Keenan JD, Gaynor BD, Porco TC, Lietman TM, Martin DL. Community-level chlamydial serology for assessing trachoma elimination in trachoma-endemic Niger. PLoS Negl Trop Dis. 2019 Jan 28;13(1):e0007127. doi: 10.1371/journal.pntd.0007127. eCollection 2019 Jan. PMID 30689671
- [Derived] Keenan JD, Chin SA, Amza A, Kadri B, Nassirou B, Cevallos V, Cotter SY, Zhou Z, West SK, Bailey RL, Porco TC, Lietman TM; Rapid Elimination of Trachoma (PRET) Study Group. The Effect of Antibiotic Selection Pressure on the Nasopharyngeal Macrolide Resistome: A Cluster-randomized Trial. Clin Infect Dis. 2018 Nov 13;67(11):1736-1742. doi: 10.1093/cid/ciy339. PMID 29897440
- [Derived] O'Brien KS, Cotter SY, Amza A, Kadri B, Nassirou B, Stoller NE, Zhou Z, West SK, Bailey RL, Keenan JD, Porco TC, Lietman TM. Childhood Mortality After Mass Distribution of Azithromycin: A Secondary Analysis of the PRET Cluster-randomized Trial in Niger. Pediatr Infect Dis J. 2018 Nov;37(11):1082-1086. doi: 10.1097/INF.0000000000001992. PMID 29561511
- [Derived] Oldenburg CE, Amza A, Kadri B, Nassirou B, Cotter SY, Stoller NE, West SK, Bailey RL, Porco TC, Gaynor BD, Keenan JD, Lietman TM. Comparison of Mass Azithromycin Coverage Targets of Children in Niger: A Cluster-Randomized Trachoma Trial. Am J Trop Med Hyg. 2018 Feb;98(2):389-395. doi: 10.4269/ajtmh.17-0501. Epub 2017 Dec 14. PMID 29260659
- [Derived] Oldenburg CE, Amza A, Kadri B, Nassirou B, Cotter SY, Stoller NE, West SK, Bailey RL, Porco TC, Keenan JD, Lietman TM, Gaynor BD. Annual Versus Biannual Mass Azithromycin Distribution and Malaria Parasitemia During the Peak Transmission Season Among Children in Niger. Pediatr Infect Dis J. 2018 Jun;37(6):506-510. doi: 10.1097/INF.0000000000001813. PMID 29088030
- [Derived] Amza A, Kadri B, Nassirou B, Cotter SY, Stoller NE, West SK, Bailey RL, Porco TC, Gaynor BD, Keenan JD, Lietman TM, Oldenburg CE. Effectiveness of expanding annual mass azithromycin distribution treatment coverage for trachoma in Niger: a cluster randomised trial. Br J Ophthalmol. 2018 May;102(5):680-686. doi: 10.1136/bjophthalmol-2017-310916. Epub 2017 Sep 11. PMID 28893761
- [Derived] Bojang E, Jafali J, Perreten V, Hart J, Harding-Esch EM, Sillah A, Mabey DC, Holland MJ, Bailey RL, Roca A, Burr SE. Short-term increase in prevalence of nasopharyngeal carriage of macrolide-resistant Staphylococcus aureus following mass drug administration with azithromycin for trachoma control. BMC Microbiol. 2017 Mar 28;17(1):75. doi: 10.1186/s12866-017-0982-x. PMID 28351345
- [Derived] Amza A, Kadri B, Nassirou B, Cotter SY, Stoller NE, Zhou Z, Bailey RL, Mabey DC, Porco TC, Keenan JD, Gaynor BD, West SK, Lietman TM. A Cluster-Randomized Trial to Assess the Efficacy of Targeting Trachoma Treatment to Children. Clin Infect Dis. 2017 Mar 15;64(6):743-750. doi: 10.1093/cid/ciw810. PMID 27956455
- [Derived] Liu F, Porco TC, Amza A, Kadri B, Nassirou B, West SK, Bailey RL, Keenan JD, Lietman TM. Short-term forecasting of the prevalence of clinical trachoma: utility of including delayed recovery and tests for infection. Parasit Vectors. 2015 Oct 22;8:535. doi: 10.1186/s13071-015-1115-8. PMID 26489933
- [Derived] Liu F, Porco TC, Amza A, Kadri B, Nassirou B, West SK, Bailey RL, Keenan JD, Solomon AW, Emerson PM, Gambhir M, Lietman TM. Short-term Forecasting of the Prevalence of Trachoma: Expert Opinion, Statistical Regression, versus Transmission Models. PLoS Negl Trop Dis. 2015 Aug 24;9(8):e0004000. doi: 10.1371/journal.pntd.0004000. eCollection 2015 Aug. PMID 26302380
- [Derived] Burr SE, Hart J, Edwards T, Harding-Esch EM, Holland MJ, Mabey DC, Sillah A, Bailey RL. Anthropometric indices of Gambian children after one or three annual rounds of mass drug administration with azithromycin for trachoma control. BMC Public Health. 2014 Nov 18;14:1176. doi: 10.1186/1471-2458-14-1176. PMID 25407464
- [Derived] Gaynor BD, Amza A, Gebresailassie S, Kadri B, Nassirou B, Stoller NE, Yu SN, Cuddapah PA, Keenan JD, Lietman TM. Importance of including borderline cases in trachoma grader certification. Am J Trop Med Hyg. 2014 Sep;91(3):577-9. doi: 10.4269/ajtmh.13-0658. Epub 2014 Jul 7. PMID 25002297
- [Derived] Hart JD, Edwards T, Burr SE, Harding-Esch EM, Takaoka K, Holland MJ, Sillah A, Mabey DC, Bailey RL. Effect of azithromycin mass drug administration for trachoma on spleen rates in Gambian children. Trop Med Int Health. 2014 Feb;19(2):207-11. doi: 10.1111/tmi.12234. Epub 2014 Jan 17. PMID 24433194
- [Derived] Harding-Esch EM, Sillah A, Edwards T, Burr SE, Hart JD, Joof H, Laye M, Makalo P, Manjang A, Molina S, Sarr-Sissoho I, Quinn TC, Lietman T, Holland MJ, Mabey D, West SK, Bailey R; Partnership for Rapid Elimination of Trachoma (PRET) study group. Mass treatment with azithromycin for trachoma: when is one round enough? Results from the PRET Trial in the Gambia. PLoS Negl Trop Dis. 2013 Jun 13;7(6):e2115. doi: 10.1371/journal.pntd.0002115. Print 2013. PMID 23785525
- [Derived] Yohannan J, Munoz B, Mkocha H, Gaydos CA, Bailey R, Lietman TA, Quinn T, West SK. Can we stop mass drug administration prior to 3 annual rounds in communities with low prevalence of trachoma?: PRET Ziada trial results. JAMA Ophthalmol. 2013 Apr;131(4):431-6. doi: 10.1001/jamaophthalmol.2013.2356. PMID 23392481
- [Derived] Amza A, Kadri B, Nassirou B, Yu SN, Stoller NE, Bhosai SJ, Zhou Z, McCulloch CE, West SK, Bailey RL, Keenan JD, Lietman TM, Gaynor BD. The easiest children to reach are most likely to be infected with ocular Chlamydia trachomatis in trachoma endemic areas of Niger. PLoS Negl Trop Dis. 2013;7(1):e1983. doi: 10.1371/journal.pntd.0001983. Epub 2013 Jan 10. PMID 23326612
- [Derived] Amza A, Kadri B, Nassirou B, Stoller NE, Yu SN, Zhou Z, Chin S, West SK, Bailey RL, Mabey DC, Keenan JD, Porco TC, Lietman TM, Gaynor BD; PRET Partnership. Community risk factors for ocular Chlamydia infection in Niger: pre-treatment results from a cluster-randomized trachoma trial. PLoS Negl Trop Dis. 2012;6(4):e1586. doi: 10.1371/journal.pntd.0001586. Epub 2012 Apr 24. PMID 22545165
- [Derived] Harding-Esch EM, Edwards T, Mkocha H, Munoz B, Holland MJ, Burr SE, Sillah A, Gaydos CA, Stare D, Mabey DC, Bailey RL, West SK; PRET Partnership. Trachoma prevalence and associated risk factors in the gambia and Tanzania: baseline results of a cluster randomised controlled trial. PLoS Negl Trop Dis. 2010 Nov 2;4(11):e861. doi: 10.1371/journal.pntd.0000861. PMID 21072224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited communities with trachoma rates 20 % or higher from 3 countries - Tanzania, Gambia and Niger.
  Protocol Enrollment refers to the number of communities, not the number of participants enrolled.
  The final analysis was done at community level.
Units Other Than Participants: community
Groups:
- ≥90% Coverage With Azithromycin , Treatment Based; 80%-89% Coverage With Azithromycin : Treatment Based: Treatment to be administered at baseline then continued yearly if trachoma prevalence is greater than 5%
  In Niger, treatment will be every 6-months for children ages twelve and under.
  Azithromycin: Comparison of coverage levels at baseline treatment followed by annual treatment if prevalence of trachoma is >5%. In Niger, there will be a comparison of coverage levels in everyone versus in children ages twelve and under who are treated every 6-months.
Period: At Baseline
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coverage With Azithromycin , Treatment Based | 80%-89% Coverage With Azithromycin : Treatment Based
Started | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis)
Niger | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis)
Gambia | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis)
Tanzania | NA; 8 community (the trial was conducted at community level and data reported per community basis) | NA; 8 community (the trial was conducted at community level and data reported per community basis) | NA; 8 community (the trial was conducted at community level and data reported per community basis) | NA; 8 community (the trial was conducted at community level and data reported per community basis)
Completed | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis) | NA; 32 community (the trial was conducted at community level and data reported per community basis)
Not Completed | NA; 0 community | NA; 0 community | NA; 0 community | NA; 0 community
Period: At 3 Years
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coverage With Azithromycin , Treatment Based | 80%-89% Coverage With Azithromycin : Treatment Based
Started | NA; 40 community (In Tanzania, units in treatment arm analyzed with antibiotic arm as tf rate was not <5% by 18 months the trial was conducted at community level and data reported per community basis) | NA; 40 community (In Tanzania, units in treatment arm analyzed with antibiotic arm as tf rate was not <5% by 18 months the trial was conducted at community level and data reported per community basis) | NA; 24 community (In Tanzania, units in treatment arm analyzed with antibiotic arm as tf rate was not <5% by 18 months the trial was conducted at community level and data reported per community basis) | NA; 24 community (In Tanzania, units in treatment arm analyzed with antibiotic arm as tf rate was not <5% by 18 months the trial was conducted at community level and data reported per community basis)
Niger | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis)
Gambia | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis) | NA; 12 community (the trial was conducted at community level and data reported per community basis)
Tanzania | NA; 16 community (the trial was conducted at community level and data reported per community basis) | NA; 16 community (the trial was conducted at community level and data reported per community basis) | NA; 0 community (the trial was conducted at community level and data reported per community basis) | NA; 0 community (the trial was conducted at community level and data reported per community basis)
Completed | NA; 40 community (the trial was conducted at community level and data reported per community basis) | NA; 40 community (the trial was conducted at community level and data reported per community basis) | NA; 24 community (the trial was conducted at community level and data reported per community basis) | NA; 24 community (the trial was conducted at community level and data reported per community basis)
Not Completed | NA; 0 community | NA; 0 community | NA; 0 community | NA; 0 community

BASELINE CHARACTERISTICS:
Population: For the final analysis the main effect of stop rule was not considered in Tanzania since no communities had prevalence < 5%.Only the main effect of coverage was analyzed there.
  In Gambia and Niger stop rule was applied and analyzed along with the main effect of coverage.
Units Other Than Participants: community
Groups:
- Total: Total of all reporting groups
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coverage With Azithromycin , Treatment Based | 80%-89% Coverage With Azithromycin : Treatment Based | Total
Number analyzed (Participants) | NA | NA | NA | NA | 0
Number analyzed (community) | 40 | 40 | 24 | 24 | 128
Age, Customized [Count of Units; unit: community] — Population: We collected and analyzed data at community level.Age was not part of final analysis.
  community
    number analyzed (Participants) | NA | NA | NA | NA | NA
    Age not analyzed | NA — We collected and analyzed data at community level.Age was not part of final analysis. | NA — We collected and analyzed data at community level.Age was not part of final analysis. | NA — We collected and analyzed data at community level.Age was not part of final analysis. | NA — We collected and analyzed data at community level.Age was not part of final analysis. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Count of Units; unit: community] — Population: We collected and analyzed data at community level.Sex/Gender was not part of final analysis.
  community
    number analyzed (Participants) | NA | NA | NA | NA | NA
    Sex/Gender not analyzed | NA — We analyzed the data on community level. Gender was not part of final analyses | NA — We analyzed the data on community level. Gender was not part of final analyses | NA — We analyzed the data on community level. Gender was not part of final analyses | NA — We analyzed the data on community level. Gender was not part of final analyses | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: community] — Population: We collected and analyzed data at community level.
  community
    number analyzed (Participants) | NA | NA | NA | NA | NA
    Tanzania | 16 | 16 | 0 | 0 | 32
    Gambia | 12 | 12 | 12 | 12 | 48
    Niger | 12 | 12 | 12 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Community Prevalence of Trachoma and Ocular C. Trachomatis (CT) Infection at Baseline
Description: Mass drug administration (MDA) with azithromycin or topical tetracycline is recommended by World Health Organization (WHO) for 3 years in districts where the prevalence of trachoma is>=10 % in children aged 1-9 years.
  The prevalence of trachoma (TF) was measured using the Simplified WHO Grading System. Both eyelids were everted and tarsal conjunctiva graded for signs of clinical trachoma. Ocular photographs of right eye were taken on random samples of sentinel children to determine the drift in grading over time. To detect CT infection, an ocular swab of the right eye using a Dacron swab was collected from the sentinel kids. The swab was stored dry, and frozen until shipped and processed in the laboratory. Air control swabs were also taken to test for field and laboratory contamination.
Time Frame: At baseline
Population: At baseline 8 communities were randomized to each arm in Tanzania, 12 communities were randomized to each arm in Gambia and Niger.
  Stop rule could not be applied in Tanzania.Communities in stop arm were moved to ≥90% coverage or 80%-89% coverage with azithromycin target arm and only main effect of coverage was analyzed in Tanzania.
Measure: Mean (Standard Deviation); unit: community
Units Other Than Participants: community
Groups:
- ≥90% Coveage With Azithromycin , Treatment Based; 80%-89% Coverage With Azithromycin : Treatment Based: Treatment to be administered at baseline then continued yearly if trachoma prevalence is greater than 5%
  In Niger, treatment will be every 6-months for children ages twelve and under.
  Azithromycin: Comparison of coverage levels at baseline treatment followed by annual treatment if prevalence of trachoma is >5%. In Niger, there will be a comparison of coverage levels in everyone versus in children ages twelve and under who are treated every 6-months.
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coveage With Azithromycin , Treatment Based | 80%-89% Coverage With Azithromycin : Treatment Based
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (community) | 40 | 40 | 24 | 24
community
  Prevalence of trachoma in Tanzania at baseline: number analyzed (community) | 8 | 8 | 8 | 8
  Prevalence of trachoma in Tanzania at baseline | 30.7 (16.3) | 30.3 (13.5) | 31.1 (9.5) | 30.5 (10.4)
  C.trachomatis infection in Tanzania at baseline: number analyzed (community) | 8 | 8 | 8 | 8
  C.trachomatis infection in Tanzania at baseline | 24.6 (12.4) | 17.8 (10.3) | 23.0 (11.2) | 22.4 (23.3)
  prevalence of trachoma in Gambia at baseline: number analyzed (community) | 12 | 12 | 12 | 12
  prevalence of trachoma in Gambia at baseline | 7.4 (26.1) | 5.6 (23.1) | 6.2 (24.1) | 6.1 (23.8)
  C.trachomatis infection in Gambia at baseline: number analyzed (community) | 12 | 12 | 12 | 12
  C.trachomatis infection in Gambia at baseline | 0.9 (9.9) | 0.7 (8.6) | 1.2 (10.8) | 0.2 (2.9)
  prevalence of trachoma in Niger at baseline: number analyzed (community) | 12 | 12 | 12 | 12
  prevalence of trachoma in Niger at baseline | 28.4 (13.9) | 27.0 (17.3) | 23.9 (12.0) | 24.7 (13.0)
  C.trachomatis infection in Niger at baseline: number analyzed (community) | 12 | 12 | 12 | 12
  C.trachomatis infection in Niger at baseline | 21.9 (16.7) | 20.5 (16.8) | 15.6 (8.8) | 24.9 (14.1)

2. Primary Outcome: Community Prevalence of Trachoma and Ocular C. Trachomatis (CT) Infection at 36 Months
Description: 100 random sentinel children aged 0- 5 years per community were to be examined for prevalence of trachoma & CT infection in Tanzania & Gambia.
  50-100 random sentinel children aged 0-5 years per community were to be examined in Niger per community for prevalence of TF and CT infection.
  Outcomes are reported at the community level because raw data could not be accessed.
  There is no way to determine how many participants were examined in each arm.
Time Frame: 3 years
Population: We analyzed and reported the results of the trial at community level.
Measure: Mean (Standard Deviation); unit: community
Units Other Than Participants: community
Groups:
- ≥90% Coveage With Azithromycin, Treatment Based; 80%-89% Coverage With Azithromycin: Treatment Based: Treatment to be administered at baseline then continued yearly if trachoma prevalence is greater than 5%
  In Niger, treatment will be every 6-months for children ages twelve and under.
  Azithromycin: Comparison of coverage levels at baseline treatment followed by annual treatment if prevalence of trachoma is >5%. In Niger, there will be a comparison of coverage levels in everyone versus in children ages twelve and under who are treated every 6-months.
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coveage With Azithromycin, Treatment Based | 80%-89% Coverage With Azithromycin: Treatment Based
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (community) | 40 | 40 | 24 | 24
community
  Prevalence of trachoma (TF) in Tanzania at 3 years: number analyzed (community) | 16 | 16 | 0 | 0
  Prevalence of trachoma (TF) in Tanzania at 3 years | 9.0 (5.9) | 6.1 (4.0) |  |
  C.trachomatis infection in Tanzania at 3 years: number analyzed (community) | 16 | 16 | 0 | 0
  C.trachomatis infection in Tanzania at 3 years | 5.4 (3.7) | 4.0 (2.7) |  |
  Prevalence of trachoma (TF) in Gambia at 3 years: number analyzed (community) | 12 | 12 | 12 | 12
  Prevalence of trachoma (TF) in Gambia at 3 years | 3.0 (17.1) | 2.3 (14.9) | 3.2 (17.6) | 2.5 (15.7)
  C.trachomatis infection in Gambia at 3 years: number analyzed (community) | 12 | 12 | 12 | 12
  C.trachomatis infection in Gambia at 3 years | 0.2 (4.1) | 1.0 (9.5) | 0.7 (8.2) | 0.2 (4.2)
  Prevalence of trachoma (TF) in Niger at 3 years: number analyzed (community) | 12 | 12 | 12 | 12
  Prevalence of trachoma (TF) in Niger at 3 years | 8.9 (8.8) | 7.1 (7.8) | 5.4 (3.9) | 10.1 (10.5)
  C.trachomatis infection in Niger at 3 years: number analyzed (community) | 12 | 12 | 12 | 12
  C.trachomatis infection in Niger at 3 years | 7.1 (6.8) | 4.6 (7.9) | 3.3 (3.6) | 4.4 (6.0)
Statistical Analysis 1: Comparison: ≥90% Coverage With Azithromycin Target vs 80%-89% Coverage With Azithromycin Target; This is analysis done in Tanzania: Only the main effect of coverage was analyzed.We hypothesized that increasing the coverage of MDA to greater than 90 % as monitored in children would result in more rapid decline in infection and trachoma compared to usual coverage.Here we are looking at the prevalence of infection; Test type: Superiority — Predicted prevalence was estimated in each community using the baseline observed prevalence, treatment arm & parameters estimated from square root transformed model.For each arm estimated prevalences were averaged.Difference in adjusted mean prevalence for enhanced arm and standard arm was calculated.For confidence intervals for adjusted difference,steps 1 to 4 for 1000 bootstrap samples were repeated.Median of adjusted mean differences, corresponding 2.5 % & 97.5 % percentiles were reported; p = 0.22, Regression, Linear; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-1 to 3.8]
Statistical Analysis 2: Comparison: 80%-89% Coverage With Azithromycin Target; This is the analysis done in Tanzania: Only the main effect of coverage was analyzed.We hypothesized that increasing the coverage of MDA to greater than 90 % as monitored in children would result in more rapid decline in infection and trachoma compared to usual coverage. Here we are looking at the prevalence of trachoma; Test type: Superiority — For each community using the baseline observed prevalence, treatment arm and parameters estimated from square root transformed model we estimated predicted prevalence.For each arm we average estimated prevalences.The difference in the adjusted mean prevalence for enhanced arm and standard arm was then calculated.In order to derive the confidence intervals for the adjusted difference, we repeated Steps 1 to 4 for 1000 bootstrap samples.The median of the adjusted mean differences were reported; p = 0.73, Ordinary least squares linear regression; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-0.3 to 5.3]
Statistical Analysis 3: Comparison: ≥90% Coverage With Azithromycin Target vs 80%-89% Coverage With Azithromycin Target vs ≥90% Coveage With Azithromycin, Treatment Based vs 80%-89% Coverage With Azithromycin: Treatment Based; This is the statistical analysis for Niger: We hypothesized that increasing the coverage of MDA to greater than 90 % as monitored in children would result in more rapid decline in infection and trachoma compared to usual coverage.Here we are looking at the prevalence of infection; Test type: Superiority; p = 0.20, Regression, Linear; Median Difference (Final Values) = -4.6, 95% CI 2-sided [-11.1 to 1.9]
Statistical Analysis 4: Comparison: ≥90% Coverage With Azithromycin Target vs 80%-89% Coverage With Azithromycin Target vs ≥90% Coveage With Azithromycin, Treatment Based vs 80%-89% Coverage With Azithromycin: Treatment Based; This is the statistical analysis for Niger: We hypothesized that increasing the coverage of MDA to greater than 90 % as monitored in children would result in more rapid decline in infection and trachoma compared to usual coverage.Here we are looking at the prevalence of trachoma; Test type: Superiority; p = 0.60, Regression, Linear; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-7.7 to 12.5]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Mass drug administration was done for all the communities in each branch. Adverse events were planned to be collected per community per arm.
  No adverse event was reported in any community in all three countries.
Arm/Group | ≥90% Coverage With Azithromycin Target | 80%-89% Coverage With Azithromycin Target | ≥90% Coverage With Azithromycin , Treatment Based | 80%-89% Coverage With Azithromycin : Treatment Based
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No